CLINICAL TRIAL: NCT02011464
Title: Evaluation of the Efficacy of Exparel Delivered Into the Posterior Capsule During Knee Replacement
Brief Title: Evaluation Exparel Delivered in Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-11-02
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exparel infiltration (Experimental): Exparel infiltrated into the posterior compartment of the knee
  Interventions: Drug: Exparel
- Control (Placebo Comparator): Saline infiltrated into posterior compartment
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Exparel — Exparel is infiltrated into posterior compartment for pain control
  Other Names: Bupivacaine
  Arms: Exparel infiltration
Other: Saline — Saline is infiltrated into posterior compartment for control
  Arms: Control

SUMMARY:
Pain control after knee replacement requires analgesia to both the top (anterior) and bottom (posterior) portion of the the knee. Presently we use a nerve block for the anterior portion. The investigators want to to examine if giving Exparel into the posterior portion will give better pain relief.

Hypothesis: There is no difference in, the use of analgesics or the length and quality of analgesia and no decrease in the time to be able to accomplish simple to complex knee movements using Exparel infiltration when compared to controls.

DETAILED DESCRIPTION:
Objectives:

1. Is to assess the efficacy of pain control of Exparel vs. controls when injected into the posterior capsular space after total knee arthroplasty
2. Asses the opioid use after Exparel vs. controls
3. Asses the time to simple and complex knee movement and ambulation.
4. The safety of Exparel will be assessed by the occurrence of all postsurgical adverse events and serious adverse events through Day 30.

Methods:

After institutional review board (IRB) approval, 20 subjects will be consented to participate in the study. The study includes subjects undergoing total knee arthroplasty either under general or spinal anesthesia. This study will include men and women (18 - 75 years) who have American Society of Anesthesiologist physical classification status 1 - 3 and underwent total knee arthroplasty.

Subjects will be divided into two groups, Group A (control) to receive 20ml of saline while Group B (study) to receive 20ml of liposomal bupivacaine into the posterior capsular space during total knee arthroplasty. Patients from both groups will receive a femoral nerve block with catheter placement for continuous infusion of local anesthetic. All subjects will have access to rescue analgesics after surgery. Multimodal analgesia will supplement pain as per standard care by the anesthesia team. Tylenol Orally 1g three times daily (not to exceed 4g in 24hrs), oxycontin 10mg orally, twice/day, Celebrex 200 mg orally once a day and Percocet 5/325 prn will serve as this multimodal approach. The time, day and number of requests for break through (additional) analgesia will be noted by both anesthesia team and primary care team. Pain scores will be assessed using a 0 - 10 numeric scale. Pain will be assessed for the following intervals: hospital arrival, post anesthesia care unit (PACU) arrival, 2, 4, 8, 12, 24, 48, 72, hours later and after hospital discharge 10 +/- 5 days after the block. Pain inquiries will assess both posterior and anterior aspects of the knee. Pain at rest and for simple leg movements (knee extension, straight leg raise) to fully ambulatory will be noted. These assessments will be made in conjunction with rehabilitation and physical therapy specialists.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years inclusive and American Society of Anesthesiologist physical status 1-3
* Patients undergoing knee replacement (total knee arthroplasty)
* Subjects must be physically and mentally able to participate in the study and complete all study assessments.
* Subjects must be able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the proposed components of infiltration into the posterior capsule of the knee.

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics
* Any subject whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful performance of a appropriate Exparel infiltration into the posterior capsule of the knee.
* Any subject who in the opinion of the Investigator, might be harmed or be a poor candidate for participation in the study.
* Any subject, who in the opinion of the Investigator, is on chronic pain medicine (opioids), including large doses of non-steroidal anti-inflammatory drugs s.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.
* History of pre-existing neurological disorders/neuropathy
* Morbid Obesity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piyush Gupta, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Exparel Inflitration: Exparel infiltrated into the posterior compartment of the knee
- Control: Saline infiltrated into posterior compartment of the knee
Period: Overall Study
Arm/Group | Exparel Inflitration | Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel Inflitration | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] — Males and females between the ages 18 and 75 years old
  years | 66.1 (4.7) | 62.8 (6.0) | 64.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Subjective Pain
Description: Subject reported post-surgical pain using the visual analog scale (VAS) during the hospital stay and after discharge. This is a 0-10 point numeric rating scale where 0 is no pain and 10 is the highest level of pain.
Time Frame: 72 hours post-operative
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exparel Group/Average Pain Scores at 4 Hours; Exparel Group/Average Pain Scores at 8 Hours; Control Group/Average Pain Scores at 8 Hours: Pain scores using the Number Rating Scale (NRS) from 0 - 10
- Control Group/Average Pain Scores at 4 Hours; Exparel Group/Average Pain Scores at 12 Hours; Control Group/Average Pain Scores at 12 Hours; Exparel Group/Average Pain Scores at 24 Hours; Control Group/Average Pain Scores at 24 Hours; Exparel Group/Average Pain Scores at 48 Hours; Control Group/Average Pain Scores at 48 Hours; Exparel Group/Average Pain Scores at 72 Hours; Control Group/Average Pain Scores at 72 Hours: Pain scores using the Numeric Rating Scale (NRS) 0 - 10
Arm/Group | Exparel Group/Average Pain Scores at 4 Hours | Control Group/Average Pain Scores at 4 Hours | Exparel Group/Average Pain Scores at 8 Hours | Control Group/Average Pain Scores at 8 Hours | Exparel Group/Average Pain Scores at 12 Hours | Control Group/Average Pain Scores at 12 Hours | Exparel Group/Average Pain Scores at 24 Hours | Control Group/Average Pain Scores at 24 Hours | Exparel Group/Average Pain Scores at 48 Hours | Control Group/Average Pain Scores at 48 Hours | Exparel Group/Average Pain Scores at 72 Hours | Control Group/Average Pain Scores at 72 Hours
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
units on a scale | 3.80 (3.26) | 4.00 (2.75) | 3.44 (3.61) | 5.30 (3.02) | 3.50 (3.25) | 3.90 (2.47) | 3.80 (3.52) | 4.20 (2.82) | 2.60 (2.46) | 3.50 (2.95) | 3.00 (3.16) | 3.70 (3.50)

2. Secondary Outcome: Post-operative Narcotic Use
Description: Average postoperative narcotics administered in total milligrams of morphine equivalents
Time Frame: 72 hours post-operative
Measure: Mean (Standard Deviation); unit: mgs
Arm/Group | Exparel Inflitration | Control
Number analyzed (Participants) | 10 | 10
mgs | 4.31 (2.40) | 5.75 (3.63)

3. Other Pre Specified Outcome: Side Effects of Analgesia
Description: Secondary end points will include the incidence of opioid related side effects (nausea, vomiting, pruritis, constipation, respiratory depression, and hypoxia) and hemodynamic perturbations related to pain
Time Frame: 72 hours post-operative
Population: Number of patients with opioid related side effects (nausea, vomiting, pruritis, constipation, respiratory depression, and hypoxia) and hemodynamic perturbations related to pain
Measure: Number; unit: participants
Arm/Group | Exparel Inflitration | Control
Number analyzed (Participants) | 10 | 10
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 72 hours post-operative
Arm/Group | Exparel Inflitration | Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No